CLINICAL TRIAL: NCT06127485
Title: Effects of Neuropilates on Rehabilitation Programs for Chronic Stroke: A Randomized Clinical Trial
Brief Title: Effects of Neuropilates on Rehabilitation Programs for Chronic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Sara Garcia Bravo, PhD Physiotherapist, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3006202326123
Record Dates: First submitted 2023-10-28; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Stroke; Occupational Therapy; Physiotherapy
MeSH Terms: conditions — Stroke | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The treatment received is a combination of physiotherapy and conventional occupational therapy sessions two days a week, with a duration of 60 minutes divided into 30 minutes of physiotherapy and 30 minutes of occupational therapy.
  Interventions: Procedure: Occupational Therapy and Physiotherapy conventional
- Experimental Group (Experimental): The experimental group received 60 minutes of conventional rehabilitation combined with the Pilates Method, divided into 20 minutes of physiotherapy, 20 minutes of occupational therapy and 20 minutes of Pilates Method.
  Interventions: Procedure: Neuropilates+occupational therapy and physiotherapy conventional

INTERVENTIONS:
Procedure: Neuropilates+occupational therapy and physiotherapy conventional — Participants assigned to the experimental group received 60 minutes of conventional rehabilitation combined with the Pilates Method, divided into 20 minutes of physical therapy, 20 minutes of occupational therapy and 20 minutes of Pilates Method. Pilates routines will be performed on a mat through the practice of Pilates activation exercises. Each participant will be given the necessary adaptations of each exercise according to their difficulties/disabilities.
  Arms: Experimental Group
Procedure: Occupational Therapy and Physiotherapy conventional — Conventional physical therapy in both groups will include stretching techniques and muscle activation of the lower limb and gait reeducation. Conventional occupational therapy will include stretching techniques and muscle activation in the upper limb as well as training in activities of daily living and functional activities of the upper limb.
  Arms: Control group

SUMMARY:
Introduction: Cerebrovascular damage (stroke) can generate motor or cognitive sequelae, making rehabilitation (such as the Pilates method) necessary to improve autonomy and quality of life. However, there are no studies on the efficacy of the method in the recovery of the upper limb and the improvement of autonomy after stroke.

Methods: Randomized double-blind clinical trial with patients with stroke in semi-acute period, randomized into experimental group (EG) (conventional rehabilitation and Pilates) or control group (CG) (conventional rehabilitation).

After randomization and initial evaluation, the intervention will begin (2 sessions per week, 3 months). After completion, there will be post-intervention assessment, and another one at 1 month.

Intervention: The CG will receive 30 minutes of physical therapy and 30 minutes of occupational therapy. The SG will receive 20 minutes of physiotherapy, 20 minutes of occupational therapy and 20 minutes of Pilates.

Assessment instruments: Mean Functional Independence; Functional Range Test; Timed 'Up and Go'; Nine Hole Peg Test; Box and Block Test; Arm, Shoulder and Hand Disabilities Questionnaire; Client Satisfaction Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. present a diagnosis of ischemic or hemorrhagic stroke with a minimum evolution of 3 months;
2. be over 18 years of age;
3. regularly attend rehabilitation treatment at the Physiocare Madrid center;
4. present moderate functional problems (score greater than 65 on the Barthel Index);
5. not present moderate cognitive impairment (Mini Mental State Examination less than 18 points);
6. not present nasogastric tubes;
7. accept to participate voluntarily in the study and sign the informed consent form;
8. be able to participate in the study and sign the informed consent form.

Exclusion Criteria:

1. time of evolution of less than 3 months;
2. other conditions of the central nervous system (tumors, anoxia, cranioencephalic trauma, etc.);
3. cardiorespiratory or neurodegenerative disorders, severe brain damage or a score of 6 or higher on the Reisberg Deterioration Scale (GDS);
4. a severely impaired level of consciousness or a score of 8 or lower on the Glasgow Coma Scale (GCS);
5. receiving other complementary rehabilitative therapy;
6. a severe deterioration in the level of consciousness or a score of 8 or lower on the Glasgow Coma Scale (GCS);
7. a severe deterioration in the level of consciousness or a score of 8 or lower on the Glasgow Coma Scale (GCS);
8. a severe deterioration in the level of consciousness or a score of 8 or lower on the Glasgow Coma Scale (GCS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Functional Independance Measure (FIM) | pre-intervention (baseline); post-intervention (immediately after the intervention) and follow up (one month after the intervention)
  an instrument that measures the level of functional independence in activities of daily living. It provides information mainly on motor and cognitive performance by means of 18 items.
  items. The score ranges from 1 to 7, with a higher score corresponding to a higher level of functional independence. Administration was carried out by means of task observation and interview.
Functional Reach Test | pre-intervention (baseline); post-intervention (immediately after the intervention) and follow up (one month after the intervention)
  A test that measures the maximum distance an individual can move their center of gravity to the limits of their base of support. In a relaxed standing position, with feet at hip level, the person is instructed to make a shoulder flexion to 90 degrees and keep the hand extended. The person has to go forward as far as he/she can. The examiner records the final measurement that they manage to shift their center of gravity. Two practice trials and three recorded trials are completed, and the average is the overall mean score. This test is recorded in centimeters.
Timed 'Up and Go' (TUG) | pre-intervention (baseline); post-intervention (immediately after the intervention) and follow up (one month after the intervention)
  A test that measures the time it takes a person to get up from a chair, walk a distance of 3 meters, turn, return to the chair and sit down. This test is responsible for exploring balance and walking speed. This test is recorded in seconds
Nine Hole Peg Test | pre-intervention (baseline); post-intervention (immediately after the intervention) and follow up (one month after the intervention)
  This test measures fine manual dexterity. This is considered a "gold standard" to evaluate fine manual dexterity. It consists of placing a number of pins on a board with 9 holes and removing them as quickly as possible. This test records the time that the person uses with each upper limb.
Box and Block Test | pre-intervention (baseline); post-intervention (immediately after the intervention) and follow up (one month after the intervention)
  Test that measures the gross motor skills of the upper limbs. It consists of a wooden box that is divided into two halves by an axis, and consists of passing from one half to the other as many wooden blocks as possible with each upper limb, for 1 minute. In this test, the number of blocks that the person is able to pass in one minute with each upper limb is recorded.
Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) | pre-intervention (baseline); post-intervention (immediately after the intervention) and follow up (one month after the intervention)
  This test measures symptoms and some aspects of activity and participation according to the 9 domains described in the International Classification of Functioning, Disability and Health in the upper extremity. It is an easy and quick test to administer

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | post-intervention (immediately after the intervention)
  This is a self-administered questionnaire, consisting of 8 questions that evaluate the level of satisfaction in relation to the care and quality of service received, as well as the degree of fulfillment of the patient's expectations prior to the intervention. The answers are coded from 1-4, the total score of the questionnaire being 32 points, with higher values indicating greater satisfaction with the treatment received. In its adaptation to Spanish, it presents adequate psychometric properties and maintains the properties of the initial questionnaire. It is therefore suitable for evaluating satisfaction with the health service received in the Spanish population.

CONTACTS AND LOCATIONS:
Overall Officials: Sara García-Bravo, Study Director — Universidad Rey Juan Carlos
Locations (1):
- Physiocare Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No